CLINICAL TRIAL: NCT01819701
Title: L-carnitine and Coenzyme Q10 in Relation to the Oxidative Stress, Antioxidant Enzymes Activities, Inflammation, and the Risk of Coronary Artery Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SF11263
Record Dates: First submitted 2013-03-15; First posted 2013-03-27 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — LC1000 Posterior Composite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): starch
  Interventions: Other: Placebo
- LC and Coenzyme Q10 (Experimental): L-carnitine: 1000 mg/d and 2000 mg/d Coenzyme Q10: 150 mg/d and 300 mg/d
  Interventions: Dietary Supplement: LC-1000; Dietary Supplement: LC-2000; Dietary Supplement: Q10-150; Dietary Supplement: Q10-300

INTERVENTIONS:
Dietary Supplement: LC-1000 — L-carnitine 1000 mg /d
  Arms: LC and Coenzyme Q10
Dietary Supplement: LC-2000 — L-carnitine: 2000 mg/d
  Arms: LC and Coenzyme Q10
Dietary Supplement: Q10-150 — Coenzyme Q10: 150 mg/d
  Arms: LC and Coenzyme Q10
Dietary Supplement: Q10-300 — Coenzyme Q10: 300 mg/d
  Arms: LC and Coenzyme Q10
Other: Placebo
  Arms: Placebo

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of Taiwan. L-carnitine (LC) and coenzyme Q10 is recognized as lipid soluble antioxidants. The purposes of this study are going to investigate the relation of LC and coenzyme Q10 with the markers of lipid peroxidation, antioxidant enzymes activities, and the inflammatory markers in coronary artery disease (CAD) patients. The study is designed as a three-year study. The first year is an observation study. We will recruit CAD patients who are identified by cardiac catheterization as having at least 50% stenosis of one major coronary artery, and age-gender matched healthy subjects. The concentrations of LC, coenzyme Q10, lipid peroxidation markers (TBARS and ox-LDL), antioxidant enzymes activities (catalase, glutathione peroxidase, glutathione reductase, and superoxide dismutase), and inflammatory markers are going to analysis. The second year is a single-blind, single dose intervention study. CAD subjects are recruit form the first year and randomly assigned to placebo, coenzyme Q10-150 (150 mg/d), coenzyme Q10-300 (300 mg/d), LC-1000 (1000 mg/d) or LC-2000 (2000 mg/d) groups. Intervention is going to administration for three months. Fasting blood will be obtained in each month and determine the concentration of LC, coenzyme Q10, lipid peroxidation markers, antioxidant enzymes activities, and inflammatory markers after intervention. The third year is a single-blind, multiple doses intervention study. We are going to measure the CAD subjects from the second year intervention study. After three months washout period, the subjects are assigned to placebo, coenzyme Q10-150 plus LC-1000, coenzyme Q10-150 plus LC-2000, coenzyme Q10-300 plus LC-1000, and coenzyme Q10-300 plus LC-2000 groups. Intervention is going to administration for three months. Fasting blood will be obtained in each month and determine the concentration of LC, coenzyme Q10, lipid peroxidation markers, antioxidant enzymes activities, and inflammatory markers after intervention. Hopefully, the results of this study could provide information of LC and coenzyme Q10 supplementation for clinical dietitian in advising CAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coronary artery disease (CAD): CAD patients were identified as having at least 50% stenosis of one major coronary artery by cardiac catheterization or as have received percutaneous transluminal coronary angioplasty (PTCA).
* Health subjects: Subjects did not have any illnesses and a history of gastrointestinal disorder, cardiovascular disease (showed normal electrocardiogram), hypertension, hyperlipidemia, liver and renal disease, diabetes, cancer, alcoholism or other metabolic disease and exhibited normal blood biochemical values, including fasting blood glucose < 6.11 mmol/L, blood urea nitrogen (BUN) < 7.9 mmol/L, creatinine < 123.8 umol/L, alkaline phosphates < 190 U/L, glutamic oxaloacetic transaminase (GOT) < 35 U/L and glutamic pyruvate transaminase (GPT) < 45 U/L.
* Must be able to swallow tablets

Exclusion Criteria:

* age < 20 years old
* pregnancy women
* taking antioxidant vitamins supplements

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Antioxidant | 12 weeks
  Antioxidant ability measurements: lipid peroxidation markers (MDA), antioxidant enzymes activities (catalase, glutathione peroxidase, and superoxide dismutase).
Anti-inflammation | 12 weeks
  Measure inflammatory markers:hs-CRP, TNF-alpha, and IL-6.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Lee BJ, Lin JS, Lin YC, Lin PT. Effects of L-carnitine supplementation on lipid profiles in patients with coronary artery disease. Lipids Health Dis. 2016 Jun 17;15:107. doi: 10.1186/s12944-016-0277-5. PMID 27317162
- [Derived] Lee BJ, Lin JS, Lin YC, Lin PT. Effects of L-carnitine supplementation on oxidative stress and antioxidant enzymes activities in patients with coronary artery disease: a randomized, placebo-controlled trial. Nutr J. 2014 Aug 4;13:79. doi: 10.1186/1475-2891-13-79. PMID 25092108